CLINICAL TRIAL: NCT03787836
Title: Improving Individual Glycemic Response With Exercise Intensity
Acronym: INTENSITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Brunswick (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); New Brunswick Health Research Foundation (Other)
Responsible Party: Principal Investigator, Martin Senechal, Assistant Professor, University of New Brunswick
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-168
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: PreDiabetes; Diabetes Mellitus, Type 2; Exercise; Physical Activity
Keywords: Exercise Response; Interindividual Variability
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will first be randomized as controls or exercisers. All exercisers will complete a 16 week exercise program, then be randomized into two groups. The first group will increase the exercise intensity and conduct another 12 week program. The second group will continue the original program for an additional 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Controls (No Intervention): The primary purpose of the control participants are to provide a measure of variability. They will be used in our calculations of typical error to classify participants as responders or non-responders, and to quantify inter-individual variability.
- Exercisers (Maintained) (Experimental): The maintained exercise group will complete the original 16-week exercise intervention at an intensity of 4.5 metabolic equivalents (METs), and repeat the intervention for another 12-weeks following its completion.
  Interventions: Behavioral: Maintained Exercise
- Exercisers (Increased Intensity) (Experimental): The increased intensity exercise group will complete the original 16-week exercise intervention, followed by an additional 12 week intervention completed at an intensity of 6.0 METs.
  Interventions: Behavioral: Increased Intensity

INTERVENTIONS:
Behavioral: Maintained Exercise — Complete 28 weeks of aerobic exercise, with one week (following week 16) for testing.
  Week 1 - 16 Intensity: 4.5 metabolic equivalents (METs).
  Duration:
  Week 1: 80 minutes Week 2: 100 minutes Week 3: 120 minutes Week 4: 135 minutes Week 5 - 16: 150 minutes/week
  Week 17: Physiological Testing
  Week 18 - 29 Intensity: 4.5 METs Duration: 150 minutes/week
  All exercise must be completed across a minimum of two sessions per week. Sub-maximal exercise tests will be completed every 4 weeks to adjust intensity.
  Arms: Exercisers (Maintained)
Behavioral: Increased Intensity — Complete 28 weeks of aerobic exercise, with one week (following week 16) for testing.
  Week 1 - 16 Intensity: 4.5 metabolic equivalents (METs).
  Duration:
  Week 1: 80 minutes Week 2: 100 minutes Week 3: 120 minutes Week 4: 135 minutes Week 5 - 16: 150 minutes/week
  Week 17: Physiological Testing
  Week 18 - 29 Intensity: 6.0 METs Duration: 150 minutes/week
  All exercise must be completed across a minimum of two sessions per week. Sub-maximal exercise tests will be completed every 4 weeks to adjust intensity.
  Arms: Exercisers (Increased Intensity)

SUMMARY:
Large interindividual variability exists in the glycemic response to exercise program, resulting in a subset of individuals known as exercise non-responders (NRs). Increasing the intensity of an exercise intervention has been proposed as one method for rescuing NRs by producing beneficial changes. However, this theory has not been tested on NRs classified using glycemic outcomes. This study will evaluate if increasing the intensity of an exercise intervention will elicit a response within previous exercise NRs.

DETAILED DESCRIPTION:
Exercise can effectively slow the progression towards Type 2 diabetes (T2D). However, data suggest large interindividual variability exists in glycemic response to exercise, resulting in a subset of individuals known as exercise non-responders (NRs). Emerging research proposes that altering the parameters of an exercise intervention to provide a sufficient stimulus can elicit a response in those previously identified as NRs. To date, no research has attempted to rescue previously classified NRs based on glycemic outcomes by altering the parameters of an exercise intervention.

This study will implement an exercise program targeted at achieving the Canadian Physical Activity Guidelines, and calculate the number of NRs. We will then evaluate if increasing the intensity of exercise will elicit response to the treatment in the NRs.

Sixty adults living with prediabetes or T2D will be recruited into one of a control group, or an exercise group. The exercising participants will begin a 16-week exercise intervention, targeted at achieving 150 minutes of moderate to vigorous intensity (equating to 4.5 METs) aerobic physical activity per week. Following the 16-week exercise program, participants will be randomized into two groups, each completing an additional 12 weeks of exercise. The first will maintain the same time and intensity, while the other will complete the 150 minutes per week at an intensity equal to 6.0 METs. Randomization will occur in blocks in order to ensure an equal number of NRs in each group.

ELIGIBILITY:
Inclusion criteria:

1. Community-dwelling adults aged 19 years or older.
2. Currently living with prediabetes or T2DM as diagnosed by a physician and confirmed by an HbA1c value of 5.7% or above, as verified by duplicate testing.
3. Not currently partaking in a self-reported regular physical activity regimen, defined as consistent participation in running or jogging activity, attending physical activity or exercise classes on a weekly basis, or averaging 10,000 steps per day or more over the course of 7 days.

Exclusion criteria:

1. Self reported as currently diagnosed as having, or being treated for, low iron concentrations or anemia.
2. Diagnosed with any red blood cell altering condition.
3. Currently living with any cardiovascular disease which would impact the ability to safely participate in exercise training.
4. Currently prescribed any medication which would impact the ability to use a heart rate monitor to accurately track exercise intensity.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Exercise responders following initial program | Week 17
  The number of responders to the original 16-week exercise program, based on improvement in glycated hemoglobin
Exercise responders following additional exercise program | Week 30
  The number of responders following the additional 12-week exercise program, based on improvement in glycated hemoglobin

SECONDARY OUTCOMES:
Sex | Baseline
  Participant self-reported biological sex
Family history of cardiovascular disease | Baseline
  Self-reported family history of cardiovascular disease
Family history of cardiometabolic disease | Baseline
  Self-reported family history of cardiometabolic disease
Current medication use | Baseline
  Record of quantity and dose of current medications
Physical activity patterns | Baseline
  Participant self-reported physical activity patterns and daily step counts over a 7-day period.
Daily step count | Baseline
  Daily step count as recorded over a 7-day period
Body mass | Baseline, week 17 and week 30
  Body mass (kilograms)
Height | Baseline, week 17 and week 30
  Height (centimetres)
Waist circumference | Baseline, week 17 and week 30
  Waist circumference (cm)
Fat mass | Baseline, week 17 and week 30
  Fat mass (kg)
Fat free mass | Baseline, week 17 and week 30
  Fat free mass (kg)
Cardiorespiratory fitness | Baseline, week 17 and week 30
  VO2 peak
Body mass index | Baseline, week 17, week 30
  Weight (kilograms) and height (measured in centimetres and converted to metres) will be combined to report body mass index in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Martin Senechal, PhD, Principal Investigator — University of New Brunswick
Locations (1):
- University of New Brunswick, Fredericton, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hecksteden A, Pitsch W, Rosenberger F, Meyer T. Repeated testing for the assessment of individual response to exercise training. J Appl Physiol (1985). 2018 Jun 1;124(6):1567-1579. doi: 10.1152/japplphysiol.00896.2017. Epub 2018 Jan 11. PMID 29357481
- [Background] Montero D, Lundby C. Refuting the myth of non-response to exercise training: 'non-responders' do respond to higher dose of training. J Physiol. 2017 Jun 1;595(11):3377-3387. doi: 10.1113/JP273480. Epub 2017 May 14. PMID 28133739
- [Background] de Lannoy L, Clarke J, Stotz PJ, Ross R. Effects of intensity and amount of exercise on measures of insulin and glucose: Analysis of inter-individual variability. PLoS One. 2017 May 11;12(5):e0177095. doi: 10.1371/journal.pone.0177095. eCollection 2017. PMID 28493912
- [Derived] Thomson A, Paudel Y, Rioux B, Hrubeniuk T, Senechal M. Type 2 diabetes duration and irisin response after an aerobic exercise intervention: results from the INTENSITY study. Appl Physiol Nutr Metab. 2025 Jan 1;50:1-11. doi: 10.1139/apnm-2024-0533. PMID 40456183
- [Derived] Hrubeniuk TJ, Bouchard DR, Gurd BJ, Senechal M. Can non-responders be 'rescued' by increasing exercise intensity? A quasi-experimental trial of individual responses among humans living with pre-diabetes or type 2 diabetes mellitus in Canada. BMJ Open. 2021 Apr 5;11(4):e044478. doi: 10.1136/bmjopen-2020-044478. PMID 33820788